CLINICAL TRIAL: NCT06919991
Title: A Phase 1, Open-Label, Fixed-Sequence, Drug-Drug Interaction Study of Casdatifan With Itraconazole (Strong CYP3A4 Inhibitor) and Phenytoin (Strong CYP3A4 Inducer) in Healthy Adult Participants
Brief Title: Drug-Drug Interaction Study of Casdatifan in Healthy Adult Participants (ARC-29)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ARC-29
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: AB521; Casdatifan; HIF-2α; hypoxia-inducible factor 2 alpha
MeSH Terms: interventions — Itraconazole; Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Casdatifan-Itraconazole-Phenytoin (Experimental): Participants will receive casdatifan, itraconazole, and phenytoin.
  Interventions: Drug: Casdatifan; Drug: Itraconazole; Drug: Phenytoin

INTERVENTIONS:
Drug: Casdatifan — Administered as a single dose in treatment Periods 1, 2, and 3
Drug: Itraconazole — Administered as multiple doses in treatment Period 2
Drug: Phenytoin — Administered as multiple doses in treatment Period 3

SUMMARY:
The purpose of the study is to assess the effects of multiple doses of itraconazole (a strong CYP3A4 inhibitor) on single dose PK of casdatifan in healthy adults and to assess the effects of multiple doses of phenytoin (a strong CYP3A4 inducer) on single dose PK of casdatifan in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female 18-55 years of age, inclusive, at the screening visit.
* Male participants must be vasectomized
* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing based on participant self-reporting.
* BMI ≥ 18.0 and ≤ 32.0 kg/m2 and body weight ≥ 45 kg, at the screening visit
* Able to swallow multiple tablets and/or capsules.

Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
* History of asthma or chronic obstructive pulmonary disease (including childhood), clinically significant food allergies or anaphylaxis, as deemed by PI or designee.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-10-18 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Drug Concentration-Time Curve (AUC) for casdatifan | Up to 168 hours post dose for Period 1; up to 216 hours post dose for Period 2; and up to 120 hours post dose for Period 3
Maximum Concentration (Cmax) in Plasma for casdatifan | Up to 168 hours post dose for Period 1; up to 216 hours post dose for Period 2; and up to 120 hours post dose for Period 3
Time to Maximum Concentration (Tmax) in Plasma for casdatifan | Up to 168 hours post dose for Period 1; up to 216 hours post dose for Period 2; and up to 120 hours post dose for Period 3

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 26.2 weeks
Concentration observed at the end of the dosing interval (Ctrough) for itraconazole (Period 2) and phenytoin (Period 3) | Up to 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy/